CLINICAL TRIAL: NCT05580185
Title: Multicenter, Multinational, Follow-Up Clinical Trial of the Performance of RESPINOR DXT to Identify Patients at Increased Risk of Weaning Failure
Acronym: DE-RISK WF II
Status: Completed | Type: Observational
Sponsor: Respinor AS (Industry)
Collaborators: Centaur Clinical CRO (Unknown); Link Medical Research AS (Unknown)
Responsible Party: Sponsor
Other Study IDs: DXT-CS-007
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Failure
Keywords: Diaphragm ultrasound; Diaphragm function; Mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weaning failure: Defined as the failure to pass a spontaneous breathing trial or the need for reintubation or death within 48 hours after extubation
  Interventions: Device: RESPINOR DXT
- Weaning success: Defined as a successful spontaneous breathing trial and is not reintubated or dies in the first 48 hours after extubation
  Interventions: Device: RESPINOR DXT

INTERVENTIONS:
Device: RESPINOR DXT — Blinded, continuous diaphragmatic excursion measurements by DXT will be conducted during the patients' first SBT. The recording shall be initiated 15 minutes prior to the first SBT and will end 15 minutes post SBT.

SUMMARY:
The study will be a multicenter, multinational, prospective single arm blinded non-interventional follow-up study (from DXT-CS-005) to validate RESPINOR DXT's performance to identify patients at increased risk of weaning failure during the spontaneous breathing trial (SBT). Continuous diaphragmatic excursion measurements by RESPINOR DXT will be conducted during the patients' first SBT. The recording shall be initiated 15 minutes prior to the first SBT and will end 15 minutes post SBT.

All patients on mechanical ventilation in the ICU meeting the eligibility criteria shall undergo a daily screen for weaning readiness. If any of the components of the daily screen is not met, the patient will not undergo a SBT that day and continued to be screened daily. Patients passing daily screening criteria shall automatically receive an SBT.

The SBT shall last for 30-120 minutes and be performed on continuous positive airway pressure up to 5 cm H2O and pressure support up to 7 cm H2O. The SBT shall be terminated, and mechanical ventilation reinstituted at the original settings if the patient meets any of the SBT failure criteria.

A trial is considered successful, and physicians will be asked to approve extubation when the patient can breathe spontaneously for the whole trial.

As part of the clinical investigation, patients shall be continued to be screened daily until extubation, 21 days after enrollment, the performance of tracheostomy, death, or withdrawal of care. All patients shall be followed until hospital discharge or death.

DETAILED DESCRIPTION:
Weaning will be conducted by the clinician in charge of the patient, in accordance with the rules of good practice from the international consensus conference on withdrawal from MV (Boles, et al., 2007). Patients eligible for the study will perform a first spontaneous breathing trial (SBT) during which they will remain connected to the ventilator for 30-120 minutes on continuous positive airway pressure up to 5 cm H2O and pressure support up to 7 cm H2O, according to the recommendations of the international consensus conference on intensive care medicine (Boles, et al., 2007) and usual practices of the service.

During the SBT, the diaphragm excursion (DE) and respiratory rate shall be measured continuously using the investigative device, RESPINOR DXT, designed by the sponsor, RESPINOR (Oslo, Norway) for all patients.The continuous measurements shall be initiated 15 minutes prior to the SBT and last until 15 minutes post SBT. The investigator will be blinded to the DXT output. The DXT control unit will only display the signal needed to confirm good quality. During blinding mode, all quantifiable data are hidden from the screen; In the case DXT does not initiate blinding mode, the investigators shall enter this in the eCRF and report to the sponsor. In case of blinding failure, the patient will be excluded from the primary and secondary endpoint analysis (data marked as missing). Sensitivity analyses may, however, be conducted by including data pertaining to such unblinded patients. The patient can still be included in the descriptive secondary endpoints (including safety).

Additionally, information on VT and RR from the ventilator should be noted for the 2nd minute of the SBT.

The SBT will be interrupted and considered a failure in case of any of the SBT failure criteria:

* Respiratory rate > 35 breaths/min
* Increased accessory muscle activity
* SpO2 persistently below 90% on FiO2 < 0.4
* Heart rate persistently above 140 beats/min
* Systolic arterial blood pressure < 90 mmHg or > 180 mmHg
* Appearance of cyanosis or mottling
* Depressed mental status or agitation

A trial is considered successful, and physicians will be asked to approve extubation when the patient can breathe spontaneously for the whole trial. The patient may receive oxygen supplementation by nasal cannula or mask as needed.

The pathophysiology of weaning failure is often complex and multifactorial-respiratory, cardiac, and neurological problems can all cause weaning failure, especially in patients who have had prolonged stays in intensive care. It is therefore important to take a structured approach, identifying each factor and addressing it in turn. The physician will therefore log the failure criteria as well as the underlying reason for weaning failure.

Depressed mental status is one of the failure criteria of spontaneous breathing trials. A patient can have resolution of the acute phase of the disease for which the patient was intubated as well as adequate respiratory and cardiac function, but still have a depressed mental status leading to weaning failure. Depressed mental status will, in most cases, not affect the DE, and as such, DXT cannot predict patients who have weaning failure solely due to depressed mental status. Another cause for weaning failure unrelated to the DE is congestive heart failure. Consequently, if a patient has weaning failure solely due to depressed mental status or congestive heart failure, the patient will be excluded from the primary endpoint analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, defined as >=18 years of age, willing and able to give informed consent (either themselves or next of kin)
2. Have undergone invasive mechanical ventilation >= 24 hours
3. Ready to wean according to criteria (from the sixth international consensus conference on intensive care medicine):

   1. Adequate cough.
   2. Absence of excessive tracheobronchial secretion.
   3. Resolution of disease acute phase for which the patient was intubated.
   4. Clinical stability, defined as stable cardiovascular status (i.e., fC < 140 beats·min-1, systolic BP 90-160 mmHg, no or minimal vasopressors) and stable metabolic status.
   5. Adequate oxygenation, defined as SaO2 > 90% on < FIO2 0.4 (or PaO2/FIO2 > 150 mmHg) and PEEP < 8 cmH2O.
   6. Adequate pulmonary function, i.e., fR < 35 breaths·min-1.
   7. Adequate mentation, defined as no sedation or adequate mentation on sedation (or stable neurologic patient), i.e., patient awake, calm and responsive to simple orders (squeeze hand, knock the head, close the eyes), no agitation.

Exclusion Criteria:

1. Not registered with a social security system nor entitled to be.
2. Central or spinal neurological injury involving central ventilatory control.
3. Presence of a neuromuscular disease involving respiratory muscles.
4. Use of muscle-paralyzing agents within 24h before the study, except if given for intubation.
5. Known paralysis of a hemidiaphragm or suspicion of paralysis of a hemidiaphragm, defined by the radiographic evidence of elevation of a dome > 2.5 cm compared to the contralateral dome.
6. Tracheostomy.
7. Body mass index >35 kg/m2.
8. Patient with therapeutic limitation, i.e., reduced expectancy to survive, defined by a Charlson Comorbidity Index < 5%.
9. Pregnant woman or protected adult.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under invasive mechanical ventilation in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Difference in the rate of weaning failure between patients with a DE < 1.0 cm compared to those with a DE > 1.1 cm. | Second minute of the SBT
  Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.0 cm will have significantly higher rate of weaning failure compared to those with a DE > 1.1 cm. The relative risk (RelR) statistic will be used to assess the null hypothesis of equality.

SECONDARY OUTCOMES:
Difference in the rate of weaning failure with reintubation failure 72 hours and 7 days after extubation between patients with a DE <1.0 cm compared to those with a DE >1.1 cm | DE values from second minute of the SBT, follow for reintubation up to 7 days
  Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.0 cm will have significantly higher rate of weaning failure compared to those with a DE > 1.1 cm. The relative risk (RelR) statistic will be used to assess the null hypothesis of equality.
Subgroup analysis on the difference in the rate of weaning failure between patients with a DE <1.0 cm compared to those with a DE >1.1 cm, excluding COVID-19 patients. Similar subgroup analysis for COVID-19 patients. | Second minute of the SBT
  Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.0 cm will have significantly higher rate of weaning failure compared to those with a DE > 1.1 cm. The relative risk (RelR) statistic will be used to assess the null hypothesis of equality.
Subgroup analysis on the difference in the rate of weaning failure between patients with a DE < 1.0 cm compared to those with a DE > 1.1 cm, excluding patients where investigators wrongly suspected diaphragm dysfunction. | Second minute of the SBT
  Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.0 cm will have significantly higher rate of weaning failure compared to those with a DE > 1.1 cm. The relative risk (RelR) statistic will be used to assess the null hypothesis of equality.
Subgroup analysis on the difference in the rate of extubation failure between patients with a DE < 1.0 cm compared to those with a DE > 1.1 cm | Second minute of the SBT
  Extubation failure is defined as the need for reintubation or death within 48 hours after extubation. Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.0 cm will have significantly higher rate of weaning failure compared to those with a DE > 1.1 cm. The relative risk (RelR) statistic will be used to assess the null hypothesis of equality.
Difference in the rate of weaning failure between patients with a DE < 1.1 cm compared to those with a DE >= 1.1 cm on the primary endpoint and secondary endpoints 1-4. | Second minute of the SBT
  Median DE measurements taken during the second minute of the SBT will be used in the analysis. The hypothesis is that patients with DE < 1.1 cm will have significantly higher rate of weaning failure compared to those with a DE >= 1.1 cm. The relative risk (RelR) statistic will be used to assess the null hypothesis of equality.
Association between median DE measurements taken during the second minute of the SBTand duration of MV prior to the first SBT, after the SBT, and total MV time. | Second minute of the SBT
  Plots of DE values versus MV duration will be presented, together with the estimated correlation coefficient.
Association between median DE measurements taken during the second minute of the SBT and duration of ICU stay prior to the first SBT, after the SBT, and total ICU time. | Second minute of the SBT
  Plots of DE values versus ICU duration will be presented, together with the estimated correlation coefficient.
Estimate thresholds for DE to predict weaning outcomes during the SBT for the whole sample. | Second minute of the SBT
  Thresholds for continuous DE will be defined by ROC curve analysis.
Rate of wrongly diagnosed diaphragm dysfunction. | Second minute of the SBT
  Failure rates for physician assessment to DE prediction will be compared using McNemar's test

OTHER OUTCOMES:
Efficacy - number of patients with overall acceptable signal quality from predefined quality criteria and time fraction during SBT with this signal quality | Through the first SBT, an average of 30 minutes
  Will be presented in tables with counts and percentages.
Safety - Skin irritation frequency and severity | Through the first SBT, an average of 30 minutes
  with options 'no irritation', slight redness', 'red and moist tissue', 'granulation tissue', and 'infection leading to debridement'. Will be presented in tables with counts and percentages.
Time spent on achieving good sensor placement | Up to 30 minutes
  with options 0-5, 6-10 mins, 11-20 mins, 21-30 mins, > 30 mins. Will be presented in tables with counts and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Demoule, MD, Principal Investigator — Hôpital Universitaire Pitié Salpêtrière
Locations (8):
- France (7):
  - Hopital Saint-Antoine, Paris, Cedex 12
  - Hôpitaux Universitaires de Marseille - AP-HM, Marseille, Chem. Des Bourrely
  - Centre Hospitalier Universitaire de Montpellier, Montpellier, Select One...
  - CHU Angers, Angers
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - CH Saint Joseph Saint Luc, Lyon
  - Hôpital Universitaire Pitié Salpêtrière, Paris
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided